CLINICAL TRIAL: NCT07250906
Title: Evaluation of the Impact of Anterior Veneers on the Quality of Life of Children With Amelogenesis Imperfecta
Brief Title: Oral Health Related Quality of Life of Children With Amelogenesis Imperfecta
Status: Recruiting | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Yelda Kasımoğlu, Assos. Prof., Istanbul University
Other Study IDs: 2025/129
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Amelogenesis Imperfecta
Keywords: quality of life; CPQ11-14
MeSH Terms: conditions — Amelogenesis Imperfecta | interventions — Dental Veneers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Veneers — Anterior veneer treatment

SUMMARY:
This project aims to evaluate the impact of anterior veneer treatment on oral health-related quality of life in children with amelogenesis imperfecta (AI). AI is an inherited disorder that causes structural defects in enamel due to genetic abnormalities, leading to aesthetic, functional, and psychosocial challenges. Enamel defects, particularly in the anterior teeth, negatively affect patients' self-confidence and social interactions. In this study, the short-term aesthetic, functional, and psychosocial effects of veneer restorations applied to children with AI will be assessed.

This research is designed as a single-center, prospective clinical study. The study population will include pediatric patients aged 11-14 years who have been clinically and radiographically diagnosed with AI at our faculty clinic. Participants' oral health-related quality of life will be evaluated before treatment and one month after treatment using the Child Perceptions Questionnaire (CPQ11-14). Psychosocial improvement will be measured using the Rosenberg Self-Esteem Scale and the Psychosocial Impact of Dental Aesthetics Questionnaire (PIDAQ), while aesthetic satisfaction will be assessed using a Visual Analogue Scale (VAS). In addition, to objectively evaluate the participants' oral hygiene and dental health, the plaque index, gingival index, bleeding on probing index, and DMFT index will be recorded.

The data obtained are expected to demonstrate the positive impact of veneer treatment on the quality of life of children with AI, emphasizing the importance of early aesthetic rehabilitation in pediatric patients. In this respect, the study aims to provide a novel clinical and psychosocial contribution to the existing literature on the management of AI in pediatric dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy,
* Aged between 11 and 14,
* Diagnosed with Amelogenesis Imperfecta,
* Need for anterior veneers,
* Both female and male volunteers

Exclusion Criteria:

* Those with systemic diseases,
* Those with a history of allergies,
* Those not diagnosed with Amelogenesis Imperfecta,
* Those without an indication for veneers,
* Those lacking adequate cooperation skills,
* Patients younger than 11 or older than 14 years will not be included in the study.

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with amelogenesis imperfecta
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-05-16 (Estimated); Study Completion 2026-08-16 (Estimated)

PRIMARY OUTCOMES:
oral health related quality of life | 3 months
  CPQ11-14

SECONDARY OUTCOMES:
self esteem | 3 months
  Rosenberg Self-Esteem Scale
psychosocial impact of dental aesthetics | 3 months
  PIDAQ
hypersensitivity | 3 months
  Wong-Baker scale
oral hygiene | 3 months
  plaque index
gingival health | 3 months
  gingival index
gingival bleeding | 3 months
  bleeding on probing
caries status | 3 months
  DMFT

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Faculty of Dentistry, Department of Pedodontics, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No